CLINICAL TRIAL: NCT01252745
Title: An Open Label, Randomized, Balanced, Three Treatment, Parallel Design, Pharmacokinetic Study of Intranasal TBS-1 Administration to Hypogonadal Men
Brief Title: Efficacy of an Intranasal Testosterone Product
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Acerus Pharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TBS-1-2010-01
Record Dates: First submitted 2010-12-01; First posted 2010-12-03 (Estimated); Results first posted 2018-04-26 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-04

CONDITIONS: Hypogonadism
MeSH Terms: conditions — Hypogonadism | interventions — Testosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 10.0 mg of TBS-1, 4.0% T.I.D. (Experimental): TBS-1 syringes pre-filled with 125 μL 4.0% gel to deliver 5.0 mg of Testosterone per nostril (intra-nasal) given t.i.d. at 2100, 0700, and 1300 hours. (total dose 30 mg/day)
  Interventions: Drug: 10.0 mg of Testosterone, 4.0% TID
- 13.5 mg of TBS-1, 4.5% B.I.D (Experimental): TBS-1 syringes pre-filled with 150 μL 4.5% gel to deliver 6.75 mg of Testosterone per nostril (intra-nasal) given b.i.d. at 2100 and 0700 hours. (total dose 27.0 mg/day)
  Interventions: Drug: 13.5 mg of Testosterone, 4.5% B.I.D
- 11.25 mg of TBS-1, 4.5% T.I.D (Experimental): TBS-1 syringes pre-filled with 125 μL 4.5% gel to deliver 5.625 mg of Testosterone per nostril (intra-nasal) given t.i.d. at 2100, 0700, and 1300 hours. (total dose 33.75 mg/day)
  Interventions: Drug: 11.25 mg of Testosterone, 4.5% T.I.D

INTERVENTIONS:
Drug: 10.0 mg of Testosterone, 4.0% TID
  Other Names: 10.0 mg of TBS-1, 4.0% TID
  Arms: 10.0 mg of TBS-1, 4.0% T.I.D.
Drug: 13.5 mg of Testosterone, 4.5% B.I.D
  Other Names: 13.5 mg of TBS-1, 4.5% B.I.D
  Arms: 13.5 mg of TBS-1, 4.5% B.I.D
Drug: 11.25 mg of Testosterone, 4.5% T.I.D
  Other Names: 11.25 mg of TBS-1, 4.5% T.I.D
  Arms: 11.25 mg of TBS-1, 4.5% T.I.D

SUMMARY:
This clinical trial will compare the pharmacokinetic profile of testosterone after repeated intranasal administration of TBS-1 of different strengths in subjects with hypogonadism

ELIGIBILITY:
Inclusion Criteria:

* Men with primary or secondary hypogonadism and a serum morning (0900 h ± 30 minutes) testosterone levels >100 ng/dl and ≤ 300 ng/dL.
* Normal Otolaryngological nasal endoscopy examination.
* Normal prostate examination (no palpable prostatic mass), and serum PSA ≤ 4.0 ng/mL.

Exclusion Criteria:

* Current treatment with other androgens (i.e. DHEA), anabolic steroids or other sex hormones
* Treatment with Estrogens, GnRH antagonists, or Growth Hormone within previous 12 months
* History of nasal surgery, specifically turbinoplasty, septoplasty, rhinoplasty, or sinus surgery.
* History of nasal disorders (e.g. polyposis, recurrent epistaxis ( > 1 nose bleed per month, abuse of nasal decongestants) or sleep apnea.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-08; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Quality of Life Medical and Research Center, Tucson, Arizona
  - Pharmax Research Clinic Inc., Miami, Florida
  - Regional Urology LLC, Shreveport, Louisiana

RESULTS

PARTICIPANT FLOW:
Groups:
- 10.0 mg Testosterone t.i.d.: TBS-1 syringes pre-filled with 125 μL 4.0% gel to deliver 5.0 mg of Testosterone per nostril (intra-nasal) given t.i.d. at 2100, 0700, and 1300 hours. (total dose 30 mg/day)
- 13.5 mg Testosterone b.i.d.: TBS-1 syringes pre-filled with 150 μL 4.5% gel to deliver 6.75 mg of Testosterone per nostril (intra-nasal) given b.i.d. at 2100 and 0700 hours. (total dose 27.0 mg/day)
- 11.25 mg Testosterone t.i.d.: TBS-1 syringes pre-filled with 125 μL 4.5% gel to deliver 5.625 mg of Testosterone per nostril (intra-nasal) given t.i.d. at 2100, 0700, and 1300 hours. (total dose 33.75 mg/day)
Period: Overall Study
Arm/Group | 10.0 mg Testosterone t.i.d. | 13.5 mg Testosterone b.i.d. | 11.25 mg Testosterone t.i.d.
Started | 8 | 7 | 7
Completed | 8 | 7 | 7
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10.0 mg Testosterone t.i.d. | 13.5 mg Testosterone b.i.d. | 11.25 mg Testosterone t.i.d. | Total
Number analyzed (Participants) | 8 | 7 | 7 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.38 (12.55) | 53.86 (11.04) | 51.57 (9.90) | 52.59 (10.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 8 | 7 | 7 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 3 | 10
  Not Hispanic or Latino | 4 | 4 | 4 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 8 | 7 | 6 | 21
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 7 | 7 | 22

OUTCOME MEASURES:

1. Primary Outcome: Cmax of Serum Testosterone
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | 10.0 mg Testosterone t.i.d. | 13.5 mg Testosterone b.i.d. | 11.25 mg Testosterone t.i.d.
Number analyzed (Participants) | 8 | 7 | 7
ng/dL | 830 (188) | 1050 (463) | 883 (346)

2. Primary Outcome: Cavg of Serum Testosterone
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: ng/dL
Groups:
- 10.0 mg of TBS-1, 4.0% T.I.D.: TBS-1 syringes pre-filled with 125 μL 4.0% gel to deliver 5.0 mg of Testosterone per nostril (intra-nasal) given t.i.d. at 2100, 0700, and 1300 hours. (total dose 30 mg/day)
  10.0 mg of Testosterone, 4.0% TID
- 13.5 mg of TBS-1, 4.5% B.I.D: TBS-1 syringes pre-filled with 150 μL 4.5% gel to deliver 6.75 mg of Testosterone per nostril (intra-nasal) given b.i.d. at 2100 and 0700 hours. (total dose 27.0 mg/day)
  13.5 mg of Testosterone, 4.5% B.I.D
- 11.25 mg of TBS-1, 4.5% T.I.D: TBS-1 syringes pre-filled with 125 μL 4.5% gel to deliver 5.625 mg of Testosterone per nostril (intra-nasal) given t.i.d. at 2100, 0700, and 1300 hours. (total dose 33.75 mg/day)
  11.25 mg of Testosterone, 4.5% T.I.D
Arm/Group | 10.0 mg of TBS-1, 4.0% T.I.D. | 13.5 mg of TBS-1, 4.5% B.I.D | 11.25 mg of TBS-1, 4.5% T.I.D
Number analyzed (Participants) | 8 | 7 | 7
ng/dL | 413 (138) | 408 (147) | 396 (110)

3. Primary Outcome: AUC0-t of Serum Testosterone
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: ng.h/dL
Arm/Group | 10.0 mg Testosterone t.i.d. | 13.5 mg Testosterone b.i.d. | 11.25 mg Testosterone t.i.d.
Number analyzed (Participants) | 8 | 7 | 7
ng.h/dL | 9920.07 (3300.65) | 9781.39 (3532.43) | 9505.03 (2650.59)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | 10.0 mg Testosterone t.i.d. | 13.5 mg Testosterone b.i.d. | 11.25 mg Testosterone t.i.d.
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 4/8 | 2/7 | 0/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10.0 mg Testosterone t.i.d. (N=8) | 13.5 mg Testosterone b.i.d. (N=7) | 11.25 mg Testosterone t.i.d. (N=7)
Dizziness (Nervous system disorders) | 2 (2) | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Excoriation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Unrelated to Study Treatment
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Unrelated to Study Treatment
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Unrelated to the Study Treatment
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) — Unrelated to the Study Treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days